CLINICAL TRIAL: NCT04342884
Title: A Multicenter, Prospective Study of COVID-19 Using Real-Time Syndromic Surveillance, Scheduled At-home Serologic Testing, and Electronic Health Records
Brief Title: COVID-19 Community Research Partnership
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB00064912; FP00000129 (Other Grant/Funding Number: North Carolina Department of Health and Human Services); SC-75D30120C08405 (Other: Centers for Disease Control and Prevention); NCT04361123 (obsolete NCT alias)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus; COVID
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clients of Wake Forest Baptist Health (WFBH)
- Health care workers of Wake Forest Baptist Health (WFBH)

SUMMARY:
The purpose of this research is to collect information about the North Carolina community's coronavirus exposures, symptoms, and health care visits due to the virus. Participation in this study will involve completing a daily questionnaire which covers participants coronavirus illness history or symptoms, health care seeking behaviors and treatments, contact with other sick people, and for health care workers, their use of personal protective equipment.

DETAILED DESCRIPTION:
Investigators will conduct a prospective, cohort study for SARS-CoV-2 infections among clients and health care workers of Wake Forest Baptist Health (WFBH). Investigators will conduct real-time syndromic respiratory disease surveillance and, for SARS-CoV-2 infections, calculate baseline seroprevalence and seroconversion rates, hazard risks from close contacts, estimate efficacy of personal protective equipment, and assess sequelae incidence. Investigators will utilize the COVID-19 Therapeutic Learning System, an Oracle developed self-reporting data collection system that can be easily modified to address these specific questions. Over the course of the study, volunteers will report daily exposures, risk reduction behaviors, and symptoms through a secure app on their smartphone, tablet, or computer. In addition to daily syndromic surveillance, at baseline and once every month after that we will use a serologic IgM/G test kit to identify infections and reinfections in volunteers and send results to the Oracle developed database. The areas covered by this study are experiencing community spread of COVID-19 but are early enough in the epidemic to capture potentially a significant number of seroconversions over the 12 months of the study. This surveillance model will be expanded to include the clients and health workers of other medical agencies in North Carolina and in other states.

ELIGIBILITY:
Inclusion Criteria:

* All clients and health care worker of WFBH are eligible for enrollment.

Exclusion Criteria:

* Health care workers who do not receive medical services through WFBH will not be enrolled.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Investigators will seek enrollment of the clients and health care workers from diverse hospitals and clinics of WFBH.
Sampling Method: Non-Probability Sample
Enrollment: 61410 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2 infection in the general population of North Carolina | baseline
  Percent of volunteers who are 2019-nCoV Ab test positive
Seroprevalence of SARS-CoV-2 infection among health care workers of North Carolina | baseline
  Percent of volunteers who are 2019-nCoV Ab test positive

SECONDARY OUTCOMES:
Cumulative incidence of SARS-CoV-2 infection | 12 month
Monthly incidence of SARS-CoV-2 infection | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 infection by age group | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 infection by sex | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 by season | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 infection by geographic area (zip code) | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 infection by preexisting comorbidities | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 infection by COVID-2 contacts | Month 1 thru month 12
Stratified incidence of SARS-CoV-2 infection by use of personal protective equipment (PPE) by health workers | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by age group | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by sex | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by season | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by geographic area (zip code) | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by preexisting comorbidities | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by COVID-2 contacts | Month 1 thru month 12
Relative risk of SARS-CoV-2 infection by use of PPE by health workers | Month 1 thru month 12
Incidence of sequelae | Month 1 thru month 12

CONTACTS AND LOCATIONS:
Overall Officials: John W Sanders, MD, MPH&TM, Principal Investigator — Wake Forest University Health Sciences
Locations (11):
- United States (11):
  - Tulane University School of Public Health and Tropical Medicine, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Medstar Health, Columbia, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Atrium Health, Charlotte, North Carolina
  - Vidant Health, Greenville, North Carolina
  - Campbell University School of Osteopathic Medicine, Lillington, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - WakeMed Health and Hospitals, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry AA, Tjaden AH, Renteria J, Friedman-Klabanoff D, Hinkelman AN, Gibbs MA, Ahmed A, Runyon MS, Schieffelin J, Santos RP, Oberhelman R, Bott M, Correa A, Edelstein SL, Uschner D, Wierzba TF; COVID-19 Community Research Partnership. Persistence of antibody responses to COVID-19 vaccines among participants in the COVID-19 Community Research Partnership. Vaccine X. 2023 Aug 11;15:100371. doi: 10.1016/j.jvacx.2023.100371. eCollection 2023 Dec. PMID 37649617
- [Derived] Ahmed A, DeWitt ME, Dantuluri KL, Castri P, Buahin A, LaGarde WH, Weintraub WS, Rossman W, Santos RP, Gibbs M, Uschner D; COVID-19 Community Research Partnership. Characterisation of infection-induced SARS-CoV-2 seroprevalence amongst children and adolescents in North Carolina. Epidemiol Infect. 2023 Apr 3;151:e63. doi: 10.1017/S0950268823000481. PMID 37009915
- [Derived] Tjaden AH, Edelstein SL, Ahmed N, Calamari L, Dantuluri KL, Gibbs M, Hinkelman A, Mongraw-Chaffin M, Sanders JW, Saydah S, Plumb ID; COVID-19 Community Research Partnership Study Group. Association between COVID-19 and consistent mask wearing during contact with others outside the household-A nested case-control analysis, November 2020-October 2021. Influenza Other Respir Viruses. 2023 Jan;17(1):e13080. doi: 10.1111/irv.13080. Epub 2023 Jan 5. PMID 36606308
- [Derived] DeWitt ME, Tjaden AH, Herrington D, Schieffelin J, Gibbs M, Weintraub WS, Sanders JW, Edelstein SL; COVID-19 Community Research Partnership. COVID-19 Symptoms by Variant Period in the North Carolina COVID-19 Community Research Partnership, North Carolina, USA. Emerg Infect Dis. 2023 Jan;29(1):207-211. doi: 10.3201/eid2901.221111. PMID 36573634
- [Derived] Friedman-Klabanoff DJ, Tjaden AH, Santacatterina M, Munawar I, Sanders JW, Herrington DM, Wierzba TF, Berry AA; COVID-19 Community Research Partnership. Vaccine-induced seroconversion in participants in the North Carolina COVID-19 community Research Partnership. Vaccine. 2022 Oct 6;40(42):6133-6140. doi: 10.1016/j.vaccine.2022.09.021. Epub 2022 Sep 12. PMID 36117003
- [Derived] Peacock JE Jr, Herrington DM, Edelstein SL, Seals AL, Plumb ID, Saydah S, Lagarde WH, Runyon MS, Maguire PD, Correa A, Weintraub WS, Wierzba TF, Sanders JW; COVID-19 Community Research Partnership Study Group. Survey of Adherence with COVID-19 Prevention Behaviors During the 2020 Thanksgiving and Winter Holidays Among Members of the COVID-19 Community Research Partnership. J Community Health. 2022 Feb;47(1):71-78. doi: 10.1007/s10900-021-01021-z. Epub 2021 Aug 12. PMID 34383157